CLINICAL TRIAL: NCT05405660
Title: : A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Dose-ranging Study to Assess the Efficacy and Safety of CDX-0159 in Patients With Chronic Inducible Urticaria
Brief Title: A Study of CDX-0159 in Patients With Chronic Inducible Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-07; 2021-006447-95 (EudraCT Number)
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Chronic Inducible Urticaria
Keywords: CDX-0159; barzolvolimab
MeSH Terms: conditions — Chronic Inducible Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- barzolvolimab 150 mg in patients with Symptomatic Dermographism (Experimental): barzolvolimab 150 mg injection subcutaneous every 4 weeks for 20 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 300 mg in patients with Symptomatic Dermographism (Experimental): barzolvolimab 300 mg injection subcutaneous every 8 weeks for 20 weeks
  Interventions: Biological: barzolvolimab
- Placebo Comparator in patients with Symptomatic Dermographism (Placebo Comparator): Placebo injection subcutaneous every 4 weeks for 20 weeks
  Interventions: Drug: Matching Placebo
- barzolvolimab 150 mg in patients with Chronic Inducible Cold Urticaria (Experimental): barzolvolimab 150 mg injection subcutaneous every 4 weeks for 20 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 300 mg in patients with Chronic Inducible Cold Urticaria (Experimental): barzolvolimab 300 mg injection subcutaneous every 8 weeks for 20 weeks
  Interventions: Biological: barzolvolimab
- Placebo Comparator in patients with Chronic Inducible Cold Urticaria (Placebo Comparator): Placebo injection subcutaneous every 4 weeks for 20 weeks
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Biological: barzolvolimab — Subcutaneous Administration
  Other Names: CDX-0159
  Arms: barzolvolimab 150 mg in patients with Chronic Inducible Cold Urticaria; barzolvolimab 150 mg in patients with Symptomatic Dermographism; barzolvolimab 300 mg in patients with Chronic Inducible Cold Urticaria; barzolvolimab 300 mg in patients with Symptomatic Dermographism
Drug: Matching Placebo — Subcutaneous Administration
  Arms: Placebo Comparator in patients with Chronic Inducible Cold Urticaria; Placebo Comparator in patients with Symptomatic Dermographism

SUMMARY:
The purpose of this study is to assess the clinical effect, the pharmacodynamics, the safety, and the pharmacokinetics of barzolvolimab (CDX-0159) in patients with Chronic Inducible Urticaria who remain symptomatic despite the use of H1-antihistamines.

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical effect, the pharmacodynamics, the safety, and the pharmacokinetics of barzolvolimab in patients with Chronic Inducible Urticaria (Cold Urticaria [ColdU] or Symptomatic Dermographism [SD]) who remain symptomatic despite the use of H1-antihistamines.

There is a screening period of up to 4 weeks, followed by a 20-week treatment period where patients will receive either barzolvolimab 150mg, 300mg or placebo, and then a 24-week follow up period where all patients are observed.

ELIGIBILITY:
Key inclusion criteria:

1. Males and females, >/= 18 years of age.
2. Diagnosis of chronic ColdU or SD >/= 3 months.
3. Diagnosis of ColdU or SD despite the use of a stable regimen of second generation non-sedating H1-antihistamine as defined by:

   1. Recurrent pruritic wheals with or without angioedema due to ColdU or SD for >/= 6 weeks at any time prior to Visit 1 despite the use of H1-antihistamines.
   2. Must be on a stable regimen of second generation non-sedating H1-antihistamine for >/= 4 weeks prior to study treatment and agree to stay on through trial.
   3. UCT < 12 during the 14 days prior to treatment.
4. Positive provocation test

   1. for ColdU patients: developing a wheal at the test site within 10 min after using TempTest® at any temperature at both screening (Visit 1) and randomization (Visit 3)
   2. for SD patients: developing a wheal at the test site within 10 min after using FricTest® with ≥ 3 pins at both screening (Visit 1) and randomization (Visit 3)
5. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days after treatment.
6. Willing and able to complete a daily symptom electronic diary and comply with study visits.

Key exclusion criteria:

1. Women who are pregnant or nursing.
2. Active Chronic spontaneous urticaria or other forms of CIndU besides ColdU or SD that may interfere with study assessments.
3. Active, pruritic skin condition in addition to CIndU.
4. Medical condition that would cause additional risk or interfere with study procedures.
5. Known active HIV, hepatitis B or hepatitis C infection.
6. Vaccination of a live vaccine within 2 months prior to study treatment (subjects must agree to avoid vaccination during the study). Inactivated vaccines are allowed such as seasonal influenza injection or COVID-19 vaccine.
7. History of anaphylaxis

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a negative provocation test at week 12 | From baseline to week 12
  Percentage of patients with a negative provocation test for Cold Inducible Urticaria [ColdU] or Symptomatic Dermographism [SD]) at week 12
  * For ColdU patients, a negative provocation test is defined as absence of wheals at the provocation site within 10 min at ≤ 4°C after provocation using TempTest®
  * For SD patients, a negative provocation test is defined as absence of wheals at the provocation site within 10 min at 0 pins after provocation using the FricTest®

SECONDARY OUTCOMES:
Change in provocation threshold and itch for ColdU | From baseline to week 12
  Mean change from baseline to week 12 in critical temperature threshold (CTT) in patients with ColdU
  CTT is defined as threshold temperature at which wheals are triggered (highest temperature for cold), assessed at the 10-minute mark
Change in provocation threshold for SD | From baseline to week 12
  Mean change from baseline to Week 12 in Critical Friction Threshold (CFT) in patients with SD
  CFT is the threshold pin number at which wheals are triggered, assessed at the 10-minute mark
Change in worst itch reported after provocation for ColdU | From baseline to week 12
  Mean change in worst itch reported by numerical rating scale after provocation testing from baseline to week 12 in patients with ColdU
Combined patients with a negative provocation test at week 12 | From baseline to week 12
  Percentage of combined patients with a negative TempTest (ColdU) or FricTest (SD) at week 12
Change in worst itch reported after provocation for SD | From baseline to week 12
  Mean change in worst itch reported by numerical rating scale after provocation testing from baseline to week 12 in patients with SD
Change in worst itch reported after provocation in both SD and ColdU | From baseline to week 12
  Mean change in worst itch reported by numerical rating scale after provocation testing from baseline to week 12 in patients with SD and ColdU combined
Percentage of patients experiencing adverse events | From baseline to week 20
  Percentage of patients experiencing treatment-emergent adverse events (TEAE) examined by ColdU patients, SD patients and in combination. A TEAE is any untoward medical occurrence in a patient administered a study treatment.

CONTACTS AND LOCATIONS:
Locations (75):
- United States (16):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Allervie Clinical Research, Montgomery, Alabama
  - One of a Kind Clinical Research Center, LLC, Paradise Valley, Arizona
  - Little Rock Allergy & Asthma CRC, Little Rock, Arkansas
  - Kern Research, Inc, Bakersfield, California
  - Allergy & Asthma Consultants, Redwood City, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Sarasota Clinical Research, Sarasota, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - Institute for Asthma and Allergy, PC/Department of Clinical Research, Chevy Chase, Maryland
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Allergy Partners of Kerrville, Kerrville, Texas
  - Allergy Associates of Utah, Murray, Utah
- Bulgaria (6):
  - Outpatient Clinic for Individual Practice for Specialized Outpatient, Razgrad
  - Medical Center Iskar- EOOD Office of Clinical Allergology, Sofia
  - "Medical Center Ekselsior" OOD, Sofia
  - "University Multiprofile Hospital for Active Treatment 'Aleksandrovska" EAD, Clinic of Clinical Allergology, Sofia
  - Medical Center "SYNEXUS SOFIA", EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment "Prof. Dr. Stoyan Kirkovich" AD, Stara Zagora
- Estonia (2):
  - Vahlberg & Pild Clinic, Tallinn
  - East Tallin Central Hospital, Tallinn
- Georgia (4):
  - High Technology Hospital Medcenter, Batumi
  - Healthy Future, Tbilisi
  - Center of Allergy and Immunology, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (13):
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - LMU Klinikum - Klinik und Poliklinik für Dermatologie und Allergologie DASZ-Dermato-Allergologisches Studien Zentrum, München, Bavaria
  - Universitaetsklinikum Giessen u. Marburg GmbH, Marburg, Hesse
  - Elbe Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Hannover Medical University, Hanover, Lower Saxony
  - Klinikum Oldenburg gGmbH - Klinik f. Dermatologie u. Allergologie, Oldenburg, Lower Saxony
  - Universitätsklinikum Düsseldorf - Dermatologie, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen Klinikum f. Dermatologie, Venerologie u. Allergologie Hufelandstr, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster Klinik u. Poliklinik f. Dermatologie, Münster, North Rhine-Westphalia
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein - Zentrum für entzündliche Hauterkrankungen, Kiel, Schleswig-Holstein
  - Institute of Allergology IFA, Berlin
  - Universitätsklinikum Heidelberg - Dermatologie, Heidelberg
- Hungary (4):
  - Semmelweis Egyetem, ÁOK, Bőr-, Nemikórtani és Bőronkológiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ (DEKK), Bőrgyógyászati Klinika, Debrecen
  - Allergo-Derm Bakos Kft, Szolnok
  - Óbudai Egészségügyi Centrum, Zalaegerszeg
- Latvia (5):
  - Balvi and Gulbene Hospital Union, Balvi
  - Pauls Stradins Clinical University Hospital, Riga
  - "LOR" Clinic, Riga
  - Children Clinical University Hospital, Riga
  - Consilium Medicum, Riga
- Lithuania (3):
  - JSC Ausros Medicinos Centras, Kaunas
  - JSC Inlita, Vilnius
  - Center of Allergy Diagnosis and Treatment, Vilnius
- Poland (8):
  - Centrum Medyczne PLEJADY, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 w Lodzi, Lodz
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Prof. Doroty Krasowskiej, Lublin
  - Uniwersytecki Szpital Kliniczny w Opolu, Pododdział Chorób Wewnętrznych i Alergologii, Opole
  - Medicome Sp. z o.o., Oświęcim
  - Medicover Integrated Clinical Services Sp. zo.o., Torun
  - Klinika Ambroziak sp. z o.o., Warsaw
- South Africa (8):
  - Iatros International, Bloemfontein, Free State
  - WorthWhile Clinical Trials, Benoni, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Ubuntu Clinical Research, Lenasia, Gauteng
  - FCRN Clinical Trial Centre Vaal Triangle, Vereeniging, Gauteng
  - Synapta Clinical Research, Durban, KwaZulu-Natal
  - Dr PJ Sebastian, Durban, KwaZulu-Natal
  - The University of Cape Town - Lung Institute, Cape Town, Mowbray
- Spain (6):
  - HGU de Alicante, Alicante
  - Hospital Bellvitge, Barcelona
  - Hospital Vall d´ Hebron, Barcelona
  - Universidad de Navarra, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: Undecided